CLINICAL TRIAL: NCT06327360
Title: Between Beliefs and Expectations in Pulmonary Fibrosis: a Prospective Cohort Study With Mixed Methods.
Brief Title: Illness Expectations in Pulmonary Fibrosis
Acronym: CAMFP
Status: Enrolling by invitation | Type: Observational
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other); FIMARP ONLUS - FEDERAZIONE ITALIANA IPF E MALATTIE POLMONARI RARE (Unknown)
Responsible Party: Principal Investigator, Eleonora Volpato, Clinical Professor, Fondazione Don Carlo Gnocchi Onlus
Other Study IDs: FDG_ 88-16
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Pulmonary Fibrosis
Keywords: Pulmonary Fibrosis; Clinical Psychology; Rehabilitation Psychology; Illness Expectations; Illness Perceptions; Adherence to treatment
MeSH Terms: conditions — Pulmonary Fibrosis; Treatment Adherence and Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with Pulmonary Fibrosis at the Don Gnocchi Foundation (Milan): 42 patients
  Interventions: Other: Psychological questionnaires
- Patients with Pulmonary Fibrosis at the Policlinico (Milano): 42
  Interventions: Other: Psychological questionnaires
- Patients with Pulmonary Fibrosis at the FIMARP ONLUS: 46
  Interventions: Other: Psychological questionnaires

INTERVENTIONS:
Other: Psychological questionnaires — The questionnaires will be completed at the time of enrollment (T0), and at the 6- and 12-month follow-ups.

SUMMARY:
This study aims to delve into the constructs of illness beliefs and expectations among patients with Pulmonary Fibrosis, exploring how these beliefs and expectations may influence the treatment journey, including oxygen therapy, non-invasive ventilation therapy, and pharmacological treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pulmonary fibrosis
* Patients using oxygen therapy
* Patients using non-invasive ventilation
* Patients undergoing pharmacological treatment
* Patients who speak and understand the Italian language

Exclusion Criteria:

* Patients who do not provide their consent
* Patients without pulmonary fibrosis
* Patients with psychiatric disorders or cognitive impaiment
* Patients who don't speak or understand Italian language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pulmonary fibrosis, at any stage, of any gender and age
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Adherence to Pharmacological Treatment | from October 2023 to October 2025
  Types of medications taken (Pirfenidone/Nintedanib/Other); assessed as the ratio between the received daily dose (RDD) and the prescribed daily dose (PDD); also evaluated using the Medication Adherence Report Scale (MARS-5), a 5-item questionnaire.
Adherence to Oxygen Therapy | from October 2023 to October 2025
  Use of oxygen and respective quantities (liters/minute at rest and during exertion).
Adherence to Non invasive ventilation | from October 2023 to October 2025
  Use of Non-Invasive Ventilation (nighttime/daytime or both; prescribed and actual hours of usage).
Illness beliefs | from October 2023 to October 2025
  Assessed using the Brief Illness Perception Questionnaire (B-IPQ), a nine-question scale designed to rapidly assess cognitive and emotional representations of the illness.
  Assessed using the Brief Illness Perception Questionnaire (B-IPQ), a nine-question scale designed to rapidly assess cognitive and emotional representations of the illness.
Pharmacological treatment Beliefs | from October 2023 to October 2025
  Assessed using the Beliefs about Medicines Questionnaire (BMQ), a tool designed to evaluate individuals' beliefs about medications. It has been validated for use in patients with chronic illnesses and has been shown to predict treatment adherence in other groups, such as individuals with asthma.
Illness Expectations | from October 2023 to October 2025
  Specific questions formulated to assess explicit illness expectations in Pulmonary Fibrosis are proposed.
Illness Cognitions | from October 2023 to October 2025
  Illness Cognition Questionnaire (ICQ), a questionnaire assessing three ways of cognitively evaluating the stressful and adverse nature of a chronic illness: helplessness, acceptance, and perceived benefits.

SECONDARY OUTCOMES:
Socio-demographic variables | from October 2023 to October 2025
  Gender, age, smoking status, and number of cigarettes smoked per day. Additionally, factors such as family history of respiratory diseases, alcohol use (frequency), physical activity (frequency and type), level of education, marital status, onset of initial symptoms, and date of diagnosis will be considered.
Clinical and medical data | from October 2023 to October 2025
  Weight and height (for calculation of Body Mass Index, BMI); comorbidities (diabetes, hypertension, hypercholesterolemia, presence of other conditions), perceived symptoms (e.g., dyspnea, cough, chest pain, fatigue and weakness, muscle and joint pains, weight loss...). Additionally, parameters from respiratory function tests (particularly Forced Vital Capacity (FVC) and Diffusing Capacity of the Lungs for Carbon Monoxide (DLCO), arterial blood gas analysis) will be recorded. These data will be extracted from the latest available medical report and therefore from the last pulmonary visit conducted as part of routine clinical practice (please note that medical visits paid for by this project are not included).

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico di Milano, Milan
  - Don Gnocchi Foundation, Milan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Raghu G, Chen SY, Hou Q, Yeh WS, Collard HR. Incidence and prevalence of idiopathic pulmonary fibrosis in US adults 18-64 years old. Eur Respir J. 2016 Jul;48(1):179-86. doi: 10.1183/13993003.01653-2015. Epub 2016 Apr 28. PMID 27126689
- [Background] Meyer KC. Pulmonary fibrosis, part I: epidemiology, pathogenesis, and diagnosis. Expert Rev Respir Med. 2017 May;11(5):343-359. doi: 10.1080/17476348.2017.1312346. Epub 2017 Apr 10. PMID 28345383
- [Background] Wolters PJ, Blackwell TS, Eickelberg O, Loyd JE, Kaminski N, Jenkins G, Maher TM, Molina-Molina M, Noble PW, Raghu G, Richeldi L, Schwarz MI, Selman M, Wuyts WA, Schwartz DA. Time for a change: is idiopathic pulmonary fibrosis still idiopathic and only fibrotic? Lancet Respir Med. 2018 Feb;6(2):154-160. doi: 10.1016/S2213-2600(18)30007-9. PMID 29413083
- [Background] Ley B, Collard HR. Epidemiology of idiopathic pulmonary fibrosis. Clin Epidemiol. 2013 Nov 25;5:483-92. doi: 10.2147/CLEP.S54815. PMID 24348069
- [Background] Broadbent E, Petrie KJ, Main J, Weinman J. The brief illness perception questionnaire. J Psychosom Res. 2006 Jun;60(6):631-7. doi: 10.1016/j.jpsychores.2005.10.020. PMID 16731240
- [Background] Evers AW, Kraaimaat FW, van Lankveld W, Jongen PJ, Jacobs JW, Bijlsma JW. Beyond unfavorable thinking: the illness cognition questionnaire for chronic diseases. J Consult Clin Psychol. 2001 Dec;69(6):1026-36. PMID 11777106
- [Background] Agarwal P, Lin J, Muellers K, O'Conor R, Wolf M, Federman AD, Wisnivesky JP. A structural equation model of relationships of health literacy, illness and medication beliefs with medication adherence among patients with chronic obstructive pulmonary disease. Patient Educ Couns. 2021 Jun;104(6):1445-1450. doi: 10.1016/j.pec.2020.11.024. Epub 2020 Nov 25. PMID 33308880